CLINICAL TRIAL: NCT05300399
Title: MIND-the-SKIN Project: Multi-functional Innovative Digital Toolkit for the Skin Diseases in LMICs and Beyond
Brief Title: Digital Toolkit for Skin Diseases in LMICs
Acronym: MIND-the-SKIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tulane University (Other)
Collaborators: Osaka University (Other); Hope Commission International (Unknown); Institut Pasteur of Cote d'Ivoire (Other Government); Institut Raoul Follereau (Unknown); Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other); Trilobite, Ltd. (Unknown)
Responsible Party: Principal Investigator, Rie Yotsu, Associate Professor, Tulane University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-2054
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Skin Diseases
Keywords: Skin Diseases; Neglected Diseases; Teledermatology; Telemedicine; Remote Consultation
MeSH Terms: conditions — Skin Diseases; Neglected Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With mHealth app (Experimental)
  Interventions: Device: mHealth app
- Without mHealth app (No Intervention)

INTERVENTIONS:
Device: mHealth app — The local healthcare providers will be assigned to an intervention group receiving the mHealth app to be used in their daily practices or a control group.
  Arms: With mHealth app

SUMMARY:
To evaluate the early detection and effective management of skin diseases using the mHealth app in Cote d'Ivoire, a mixed-methods pilot trial will be conducted in Cote d'Ivoire. The pilot trial will consist of 3 phases: phase 1, development and improvement of the mHealth app; phase 2, pilot trial to evaluate the usability of the mHealth app for local healthcare providers in Cote d'Ivoire; and phase 3, pilot trial to evaluate the effectiveness of case detection and management of skin diseases with the mHealth app in Cote d'Ivoire. The pilot study will be implemented as a 2-arm trial with local healthcare providers and patients with skin diseases over a 3-month follow-up period.

DETAILED DESCRIPTION:
Background: The prevalence of skin diseases is extremely high in sub-Saharan Africa, among which are skin neglected tropical diseases (skin NTDs) that could lead to life-long disabilities and deformities if not diagnosed and treated early. To achieve early detection and early treatment of these skin diseases, we developed a mobile health application (mHealth app): 'eSkinHealth'.

Objective: To evaluate the early detection and effective management of skin diseases using the mHealth app in Cote d'Ivoire.

Methods: A mixed-methods pilot trial will be conducted in Cote d'Ivoire and will consist of 3 phases: phase 1, development and improvement of the mHealth app; phase 2, pilot trial to evaluate the usability of the mHealth app for local healthcare providers in Cote d'Ivoire; and phase 3, pilot trial to evaluate the effectiveness of case detection and management of skin diseases with the mHealth app in Cote d'Ivoire. The pilot study will be implemented as a 2-arm trial with local healthcare providers and patients with skin diseases over a 3-month follow-up period.

Local healthcare providers (i.e., doctors, nurses, or community health workers/volunteers) must meet all eligibility requirements to enroll in the study. Eligible local healthcare providers are; (1) 18 years or older, (2) working at primary health centers or clinics in Cote d'Ivoire, (3) able to read and speak fluent French, (4) willing to participate in the pilot study for the 3-month study duration and use a provided tablet with the eSkinHealth app if they were assigned in the intervention group, and (5) able to consent for oneself. Ineligible local healthcare providers will be defined as those who (1) are planning to leave the job at the clinics within the study period and (2) have difficulty in operating mobile devices.

Eligible patients will be defined as those are; (1) clinically suspected or diagnosed of skin NTDs (Buruli ulcer, leprosy, lymphatic filariasis, yaws, or other skin NTDs) or have other clinically diagnosed skin conditions, (2) diagnosed of concomitantly fewer than three identified skin conditions, and (3) able to consent for oneself. Ineligible patients have (1) more than three skin conditions and (2) clinically diagnosed skin conditions outside of the target site.

For phase 2, we will use a validated questionnaire, the system usability scale (SUS). The outcome measurement is an average score of SUS. The SUS consists of 10 statements with responses in the form of a five-point Likert scale (e.g., 1: strongly disagree, 5: strongly agree). We will use the French-language version of SUS. We will assess the usability at baseline, midpoint (6 weeks), and at the end of the study (12 weeks).

For phase 3, differences in case numbers diagnosed and followed up between the intervention group (with the app) and the control group (without the app) will be measured as the primary outcome of this study. We will also evaluate the effectiveness of the intervention on secondary outcomes, including engagement with the app's platform and willingness to use it. The engagement of local healthcare providers will be measured via data usage, including the frequency of visits to the platform and time spent there.

ELIGIBILITY:
Phase 2: Local healthcare providers (i.e., doctors, nurses, or community health workers/volunteers)

Inclusion Criteria:

* 18 years or older
* Working at primary health centers or clinics in Cote d'Ivoire
* Able to read and speak fluent French
* Willing to participate in the pilot study for the 3-month study duration and use a provided tablet with the eSkinHealth app if they were assigned to the intervention group
* Able to consent for oneself

Exclusion Criteria:

* Planning to leave their job at the clinics within the study period
* Difficulty operating mobile devices

Phase 3: Patients with skin diseases

Inclusion Criteria:

* Clinically suspected or diagnosed with skin NTDs (Buruli ulcer, leprosy, and yaws) or have other clinically diagnosed skin conditions
* Diagnosed of concomitantly fewer than three identified skin conditions
* Able to consent for oneself

Exclusion Criteria:

* More than three skin conditions
* Clinically diagnosed skin conditions outside of the target site

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1364 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Differences in case numbers diagnosed and followed up | 12 weeks
  Differences in case numbers diagnosed and followed up between the intervention group (with the app) and the control group (without the app) will be measured as the primary outcome of this study.

SECONDARY OUTCOMES:
Effectiveness of the app | 12 weeks
  We will assess the engagement with the app's platform and willingness to use it. The engagement of local healthcare providers will be measured via data usage, including frequency of visit to the platform and time spent there.
Usability of the app | 12 weeks
  We will assess the usability of the app at baseline, midpoint (6 weeks), and at the end of the study (12 weeks). The outcome measurement is an average score of SUS. The SUS consists of 10 statements with responses in the form of a five-point Likert scale (e.g., 1: strongly disagree, 5: strongly agree). We will use the French-language version of SUS.

CONTACTS AND LOCATIONS:
Locations (1):
- Rie Yotsu, Sinfra, Côte d’Ivoire

REFERENCES:
- [Derived] Yotsu RR, Almamy D, Vagamon B, Ugai K, Itoh S, Koffi YD, Kaloga M, Dizoe LAS, Kouadio K, Aka N, Yeboue LKG, Yao KA, Blanton RE. An mHealth App (eSkinHealth) for Detecting and Managing Skin Diseases in Resource-Limited Settings: Mixed Methods Pilot Study. JMIR Dermatol. 2023 Jun 14;6:e46295. doi: 10.2196/46295. PMID 37632977
- [Derived] Yotsu RR, Itoh S, Yao KA, Kouadio K, Ugai K, Koffi YD, Almamy D, Vagamon B, Blanton RE. The Early Detection and Case Management of Skin Diseases With an mHealth App (eSkinHealth): Protocol for a Mixed Methods Pilot Study in Cote d'Ivoire. JMIR Res Protoc. 2022 Sep 21;11(9):e39867. doi: 10.2196/39867. PMID 35922062